CLINICAL TRIAL: NCT06613321
Title: Impact of Lung Hyperinflation on the Response to Pulmonary Vasodilator Therapy in Patients with Pulmonary Hypertension (PH) Associated with Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Lung Hyperinflation and Response to Pulmonary Vasodilator Therapy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PI014
Record Dates: First submitted 2023-10-09; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Copd; Hypertension, Pulmonary; Hyperdistention
Keywords: copd; pulmonary distension; lung distension disorders; pulmonary hypertension; vasodilator therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with increased lung distension: Defined by a residual volume over total lung capacity ratio (RV/TLC ratio) above the median value of all included patients.
  Interventions: Diagnostic Test: Respiratory function tests before introduction of vasodilator therapy; Diagnostic Test: 3 month follow up evaluation of response to treatment.
- Patients without increased distension disorder: Defined by a residual volume over total lung capacity ratio (RV/TLC ratio) below the median value of all included patients.
  Interventions: Diagnostic Test: Respiratory function tests before introduction of vasodilator therapy; Diagnostic Test: 3 month follow up evaluation of response to treatment.

INTERVENTIONS:
Diagnostic Test: Respiratory function tests before introduction of vasodilator therapy — Respiratory function tests before introduction of vasodilator therapy with evaluation of the RV/TLC ratio.
Diagnostic Test: 3 month follow up evaluation of response to treatment. — Follow up of patients at least 3 months after introduction of vasodilator therapy to determine response to treatment or absence of response.

SUMMARY:
The goal of this retrospective observational study is to evaluate if lung distension disorders can be a predictive factor of bad response to vasodilator therapy in patients with pulmonary hypertension (PH) associated with chronic obstructive pulmonary disease (COPD).

The study will include all patients from the hospital, followed for pulmonary hypertension associated with COPD under vasodilator therapy between 2015 and 2021.

DETAILED DESCRIPTION:
The goal of this retrospective observational study is to evaluate if lung distension disorders can be a predictive factor of bad response to vasodilator therapy in patients with pulmonary hypertension (PH) associated with chronic obstructive pulmonary disease (COPD).

The study will include all patients from the hospital, followed for PH associated with COPD under vasodilator therapy between 2015 and 2021.

It will evaluate patients' lung hyperinflation according to the RV/TLC ratio and their response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD regardless of severity defined as a FEV1/FVC ratio less than 0.70 and the presence of a risk factor (smoke exposure with at least a 10 pack-year history, or professional exposition) diagnosed with PH according to ESC/ERS 2022 classification and in whom vasodilator therapy has been initiated

Exclusion Criteria:

* other known concomitant lung disease (interstitial lung disease, cystic lung disease, mucoviscidosis…)
* thoracic pathology such as kyphoscoliosis
* pleural effusion (unless part of pulmonary veno-occlusive disease)
* a large tumor lung mass
* EFR missing or uninterpretable because difficult to perform
* initiation of calcium channel blockers
* surgical treatment in chronic thrombo-embolic pulmonary hypertension
* no follow-up evaluation (lost to follow-up or died before reassessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with pulmonary hypertension associated with COPD undergoing vasodilator therapy at Nancy University Hospital (France) from January 1, 2015 to April 1, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 3 - 12 months
  Response to treatment is defined as an improvement of at least 30 meters in the 6-minute walk test or one NYHA functional class at the first re-evaluation performed at least 3 months after the initiation of vasodilator therapy. These criteria will be compared according to the severity of chest distension.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Chaouat, MD PhD, Principal Investigator — Université de Lorraine, Département de Pneumologie, CHRU NANCY
Locations (1):
- CHU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farkouh C, Chaouat A, Guillaumot A, Baptista BR, Chabot F, Valentin S. Pulmonary hypertension in patients with chronic obstructive pulmonary disease: Impact of lung hyperinflation on the response to pulmonary hypertension treatment. Respir Med Res. 2025 May;87:101153. doi: 10.1016/j.resmer.2024.101153. Epub 2024 Dec 18. PMID 39765128